CLINICAL TRIAL: NCT03151317
Title: Effects of a Therapeutic Education Program on Treatment Adherence Among Patients Prescribed At-home Continuous Positive Airway Pressure or At-home Non-invasive Ventilation
Brief Title: Effects of a Therapeutic Education Program on Treatment Adherence Among Patients Prescribed At-home CPAP or At-home NIV
Acronym: APARDetp
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Association pour l'Assistance et la Réhabilitation à Domicile (APARD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0077
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2017-05

CONDITIONS: Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With therapeutic education: Patients assigned to this group will have participated in a therapeutic education program.
- Without therapeutic education (control): Patients assigned to this (control) group have not had any kind of therapeutic education.

SUMMARY:
The primary objective of this study is to study the effect of therapeutic education on patient adherence for at-home continuous positive airway pressure (CPAP) or at-home non-invasive ventilation. This first study will use data already present in the Association for Home Assistance and Rehabilitation (APARD) database to compare patients who received therapeutic education with a control group who did not.

DETAILED DESCRIPTION:
The proposed study calendar refers to the beginning and completion of work on the APARD database.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have been equipped by the Association for Home Assistance and Rehabilitation (APARD) with either a continuous positive airway pressure (CPAP) device or a non-invasive ventilation (NIV) device.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of patients that have been equipped by the Association for Home Assistance and Rehabilitation (APARD) with either a continuous positive airway pressure (CPAP) device or a non-invasive ventilation (NIV) device.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Treatment adherence | a period of 28 days (retrospective study)
  Treatment adherence will be quantified as the average number of hours of device usage per night

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Molinari, PhD, Study Director — University Hospitals of Montpellier
Locations (1):
- Apard Database, Montpellier, France

REFERENCES:
- See also: APARD etp on the Open Science Framework — http://osf.io/6t9ks